CLINICAL TRIAL: NCT01107977
Title: Iyengar Yoga for Young People With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1K01AT005093 (NIH)
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iyengar yoga (Experimental)
  Interventions: Behavioral: Iyengar yoga
- Waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: Iyengar yoga — Iyengar yoga twice/week for 6 weeks
  Arms: Iyengar yoga

SUMMARY:
Irritable bowel syndrome (IBS) affects as many as 14% of high school-aged students. Symptoms include discomfort in the abdomen, along with diarrhea and/or constipation and other gastroenterological symptoms, which can significantly impact quality of life and daily functioning of patients. Emotional stress appears to exacerbate IBS symptoms suggesting that mind-body interventions reducing arousal may prove beneficial. Often symptoms can be traced to childhood and adolescence, making the early manifestation of IBS important to understand. The current study focuses on young people aged 14-26 years of age with IBS. The study will test the potential benefits of Iyengar yoga (IY) on clinical symptoms, psychospiritual functioning and visceral sensitivity. Yoga is thought to bring physical, psychological and spiritual benefits to practitioners and has been associated with reduced stress and pain. Through its focus on restoration and use of props, IY is especially designed to decrease arousal and promote psychospiritual resources in physically compromised individuals. Sixty-four IBS patients aged 14-26 will be randomly assigned to a standardized 6-week biweekly IY group-based program (1.5 hour sessions) or a wait-list usual care control group. The groups will be compared on the primary clinical outcomes of IBS symptoms, quality of life and global improvement at post-treatment and 2 month follow-up. Secondary outcomes will include visceral pain sensitivity assessed with a standardized laboratory task (water load task), and psychospiritual variables including coping, self-efficacy, mood, acceptance and mindfulness. It is hypothesized that IY will be safe and feasible: with less than 20% attrition; and the IY group will demonstrate significantly improved outcomes compared to controls, with physiological and psychospiritual mechanisms contributing to improvements; clinical treatment gains will be maintained at 2 months following yoga.

ELIGIBILITY:
Inclusion Criteria:

* Male and female youth will be eligible for the study if they meet the following criteria:

  * Age 14-26 years.
  * Diagnosis of IBS, using ROME III pediatric criteria for patients aged 14-17 years, and ROME III adult criteria for 18-26 year-olds.
  * Able and willing to give written informed assent or consent and comply with the requirements of the study protocol.
  * Ability to speak and understand English.

Exclusion Criteria:

* Any other injury, disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion that it might affect the interpretation of the results or render the patient at high risk from treatment complications.

  * Inability to comply with study and follow-up procedures.
  * Currently pregnant.
  * Previous practice of yoga within the past three months.
  * Inability to speak and understand English.
  * Plan to begin a new treatment within 2 weeks of the IYP.

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Irritable bowel symptoms | baseline (within 2 weeks of receiving intervention)
Irritable bowel symptoms | post-intervention (within 2 weeks of completing intervention)
Irritable bowel symptoms | follow up (2 months after completion of intervention)
Quality of Life | baseline (within 2 weeks of receiving intervention)
Quality of Life | post-intervention (within 2 weeks of completing intervention)
Quality of Life | follow up (2 months after completion of intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Subhadra Evans, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Pediatric Pain Program, Los Angeles, California, United States

REFERENCES:
- [Result] Evans S, Lung KC, Seidman LC, Sternlieb B, Zeltzer LK, Tsao JC. Iyengar yoga for adolescents and young adults with irritable bowel syndrome. J Pediatr Gastroenterol Nutr. 2014 Aug;59(2):244-53. doi: 10.1097/MPG.0000000000000366. PMID 25025601
- [Derived] Evans S, Cousins L, Tsao JC, Sternlieb B, Zeltzer LK. Protocol for a randomized controlled study of Iyengar yoga for youth with irritable bowel syndrome. Trials. 2011 Jan 18;12:15. doi: 10.1186/1745-6215-12-15. PMID 21244698